CLINICAL TRIAL: NCT01252732
Title: A Multicenter, Double-Blind, Randomized Study to Evaluate the Efficacy and Safety of Single-Dose IV Oritavancin Versus IV Vancomycin for the Treatment of Patients With Acute Bacterial Skin and Skin Structure Infection (SOLO II)
Brief Title: Oritavancin Versus IV Vancomycin for the Treatment of Patients With Acute Bacterial Skin and Skin Structure Infection
Acronym: SOLO II
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Melinta Therapeutics, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: TMC-ORI-10-02
Record Dates: First submitted 2010-12-01; First posted 2010-12-03 (Estimated); Results first posted 2021-04-13 (Actual); Last update posted 2021-05-05 (Actual); Status verified 2021-04

CONDITIONS: Wound Infection; Abscess; Systemic Inflammation; Cellulitis
Keywords: ABSSSI; Skin Infection; Abscess
MeSH Terms: conditions — Wound Infection; Abscess; Cellulitis | interventions — Vancomycin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Single-Dose IV Oritavancin Diphosphate (Experimental)
  Interventions: Drug: Single-Dose IV Oritavancin Diphosphate
- IV Vancomycin (Active Comparator)
  Interventions: Drug: IV Vancomycin

INTERVENTIONS:
Drug: Single-Dose IV Oritavancin Diphosphate — Intravenous oritavancin and IV placebo or IV vancomycin will be administered for a minimum of 7 days up to a maximum of 10 days.
  Arms: Single-Dose IV Oritavancin Diphosphate
Drug: IV Vancomycin — Intravenous oritavancin and IV placebo or IV vancomycin will be administered for a minimum of 7 days up to a maximum of 10 days.
  Arms: IV Vancomycin

SUMMARY:
The purpose of this Phase 3 trial is to evaluate the efficacy, safety, and tolerability of oritavancin in ABSSSIs, including those caused by MRSA and to evaluate the potential economic benefit of oritavancin administered as a single 1200 mg IV dose.

DETAILED DESCRIPTION:
This is a Phase 3, multicenter, randomized, double-blind, parallel, comparative efficacy and safety study of single-dose IV oritavancin/IV placebo versus IV vancomycin for 7 to 10 days in adults with acute bacterial skin and skin structure infection (ABSSSI) suspected or proven to be caused by Gram-positive pathogens. Approximately 960 patients will be randomized at 100 centers globally.

In addition, this study will characterize the PK and PK/PD properties of a single 1200 mg IV dose of oritavancin and evaluate the potential health economic benefits offered by this dosing strategy.

ELIGIBILITY:
Inclusion Criteria:

Subjects may be included in the study if they meet all of the following inclusion criteria:

1. Males or females ≥18 years old
2. Diagnosis of ABSSSI suspected or confirmed to be caused by a Gram-positive pathogen requiring at least 5 days of IV therapy
3. An ABSSSI includes one of the following infections Wound infections, Cellulitis/erysipelas, Major cutaneous abscess
4. ABSSSI must present with at least 2 signs and symptoms
5. Able to give informed consent and willing to comply with all required study procedures

Exclusion Criteria:

Subjects will be excluded from the study if any of the following exclusion criteria apply prior to randomization:

1. Prior systemic or topical antibacterial therapy with activity against suspected or proven Gram-positive pathogens within the preceding 14 days

   * The causative Gram-positive pathogen(s) isolated from the ABSSSI site is resistant in vitro to the antibacterial(s) that was administered with documented clinical progression, or
   * Documented failure to previous ABSSSI antibiotic therapy is available. Documentation of treatment failure must be recorded
   * Patient received a single dose of a short acting antibacterial therapy three or more days before randomization
2. Infections associated with, or in close proximity to, a prosthetic device
3. Severe sepsis or refractory shock
4. Known or suspected bacteremia at time of screening
5. ABSSSI due to or associated with any of the following:

   * Infections suspected or documented to be caused by Gram-negative pathogens -- Wound infections (surgical or traumatic) and abscesses with only Gram-negative pathogens
   * Diabetic foot infections
   * Concomitant infection at another site not including a secondary ABSSSI lesion
   * Infected burns
   * A primary infection secondary to a pre-existing skin disease with associated inflammatory changes
   * Decubitus or chronic skin ulcer, or ischemic ulcer due to peripheral vascular disease
   * Any evolving necrotizing process gangrene or infection suspected or proven to be caused by Clostridium species
   * Infections known to be caused by a Gram-positive organism with a vancomycin MIC >2 μg/mL or clinically failing prior therapy with glycopeptides
   * Catheter site infections
6. Allergy or intolerance to aztreonam or metronidazole in a patient with suspected or proven polymicrobial wound infection involving Gram-negative and/or anaerobic bacteria
7. Currently receiving chronic systemic immunosuppressive therapy
8. AIDS with CD4 count < 200 cells/mm3
9. Neutropenia
10. Significant or life-threatening condition that would confound or interfere with the assessment of the ABSSSI
11. Women who are pregnant or nursing
12. History of immune-related hypersensitivity reaction to glycopeptides
13. Patients that require anticoagulant monitoring with an aPTT
14. Contraindication to vancomycin
15. Patients unwilling to forego blood and/or blood product donation
16. Treatment with investigational medicinal product within 30 days before enrollment and for the duration of the study
17. Investigational device present, or removed <30 days before enrollment, or presence of device-related infection
18. Patients unlikely to adhere to the protocol, comply with study drug administration, or complete the clinical study
19. Severe hepatic disease
20. Presence of hyperuricemia
21. Unwilling to refrain from chronic use of any medication with antipyretic properties

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1019 (Actual)
Dates: Start 2010-12; Primary Completion 2013-06 (Actual); Study Completion 2013-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: G. Ralph Corey, MD, Principal Investigator — Duke Clinical Research Institute
Locations (1):
- Sharp Grossmont Hospital, La Mesa, California, United States

REFERENCES:
- [Derived] Corey GR, Loutit J, Moeck G, Wikler M, Dudley MN, O'Riordan W; SOLO I and SOLO II investigators. Single Intravenous Dose of Oritavancin for Treatment of Acute Skin and Skin Structure Infections Caused by Gram-Positive Bacteria: Summary of Safety Analysis from the Phase 3 SOLO Studies. Antimicrob Agents Chemother. 2018 Mar 27;62(4):e01919-17. doi: 10.1128/AAC.01919-17. Print 2018 Apr. PMID 29358292
- [Derived] Deck DH, Jordan JM, Holland TL, Fan W, Wikler MA, Sulham KA, Ralph Corey G. Single-Dose Oritavancin Treatment of Acute Bacterial Skin and Skin Structure Infections: SOLO Trial Efficacy by Eron Severity and Management Setting. Infect Dis Ther. 2016 Sep;5(3):353-61. doi: 10.1007/s40121-016-0119-9. Epub 2016 Jul 1. PMID 27370913
- [Derived] Corey GR, Good S, Jiang H, Moeck G, Wikler M, Green S, Manos P, Keech R, Singh R, Heller B, Bubnova N, O'Riordan W; SOLO II Investigators. Single-dose oritavancin versus 7-10 days of vancomycin in the treatment of gram-positive acute bacterial skin and skin structure infections: the SOLO II noninferiority study. Clin Infect Dis. 2015 Jan 15;60(2):254-62. doi: 10.1093/cid/ciu778. Epub 2014 Oct 6. PMID 25294250

RESULTS

PARTICIPANT FLOW:
Groups:
- Single-Dose 1200 mg Oritavancin: Single 1200 mg IV Dose of Oritavancin Diphosphate administered as first infusion followed by IV placebo administered twice daily for a minimum of 7 days up to a maximum of 10 days.
- Vancomycin: IV Vancomycin, 1g or 15mg/kg administered twice daily for a minimum of 7 days up to a maximum of 10 days.
Period: Overall Study
Arm/Group | Single-Dose 1200 mg Oritavancin | Vancomycin
Started | 509 (Randomized) | 510 (Randomized)
Modified Intent to Treat Population | 503 | 502
Completed | 455 | 446
Not Completed | 54 | 64

BASELINE CHARACTERISTICS:
Population: Modified Intent to Treat (mITT) population
Groups:
- Total: Total of all reporting groups
Arm/Group | Single-Dose 1200 mg Oritavancin | Vancomycin | Total
Number analyzed (Participants) | 503 | 502 | 1005
Age, Continuous [Mean (Standard Deviation); unit: years] | 45.0 (13.40) | 44.4 (14.29) | 44.7 (13.85)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 165 | 159 | 324
  Male | 338 | 343 | 681

OUTCOME MEASURES:

1. Primary Outcome: Early Clinical Response
Description: Clinical response at the ECE visit (48-72 hours following initiation of study drug administration). Early clinical response was defined as a composite outcome based on, cessation of spreading or reduction in the size of baseline lesion, absence of fever and no rescue antibiotic medication.
Time Frame: 48-72 hours after the initation of study therapy
Population: Modified intent to treat (mITT) population consisting of all patients randomized into the trial and received any study drug.
Measure: Number; unit: participants
Arm/Group | Single-Dose 1200 mg Oritavancin | Vancomycin
Number analyzed (Participants) | 503 | 502
participants
  Success | 403 | 416
  Failure | 100 | 86
Statistical Analysis 1: Comparison: Single-Dose 1200 mg Oritavancin vs Vancomycin; Test type: Non-Inferiority or Equivalence — The non-inferiority hypothesis test is a one sided hypothesis test performed at the 2.5% level of significance. If the lower limit of the two-sided 95% CI for the difference in response rates in the mITT population is greater than -10% the NI of oritavancin to vancomycin is concluded; Difference in Proportions = -2.7, 95% CI 2-sided [-7.5 to 2.0]

2. Secondary Outcome: Investigator Assessed Clinical Cure at Post Therapy Evaluation (Key Secondary Endpoint)
Description: Compared the clinical efficacy at the Post Therapy Evaluation of Oritavancin and Vancomycin based on the Investigator examination of the signs and symptoms of the primary ABSSSI; Investigator assessment of clinical cure is complete or nearly complete resolution of baseline signs and symptoms of the primary infection such that no further treatment with antibiotics is needed
Time Frame: 7 to 14 days after end of therapy
Population: as for outcome 1
Measure: Number; unit: participants
Arm/Group | Single-Dose 1200 mg Oritavancin | Vancomycin
Number analyzed (Participants) | 503 | 502
participants
  Clinical Cure | 416 | 404
  Clinical Failure | 87 | 98
Statistical Analysis 1: Comparison: Single-Dose 1200 mg Oritavancin vs Vancomycin; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 1, analysis 1]; Difference in Proportions = 2.2, 95% CI 2-sided [-2.6 to 7.0]

3. Secondary Outcome: >= 20% Reduction in Lesion Area
Description: Clinical response at the ECE visit (48-72 hours following initiation of study drug administration) based on changes in ABSSSI lesion size measurements from baseline.
Time Frame: 48-72 hours after the initation of study therapy
Population: as for outcome 1
Measure: Number; unit: participants
Arm/Group | Single-Dose 1200 mg Oritavancin | Vancomycin
Number analyzed (Participants) | 503 | 502
participants
  Success | 432 | 428
  Failure | 71 | 74
Statistical Analysis 1: Comparison: Single-Dose 1200 mg Oritavancin vs Vancomycin; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 1, analysis 1]; Difference in Proportions = 0.6, 95% CI 2-sided [-3.7 to 5.0]

ADVERSE EVENTS:
Time Frame: Begins from the time the patient provided informed consent through to the last follow up visit at 60 (+7) days.
Description: Additional Description Adverse events were analysed in the safety population consisting of all patients who received any study drug. The analysis was performed according to the actual treatment that the patient received.
Arm/Group | Single-Dose 1200 mg Oritavancin | Vancomycin
Serious Adverse Events (participants affected / at risk) | 22/503 | 23/502
Other Adverse Events (participants affected / at risk) | 272/503 | 265/502
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Single-Dose 1200 mg Oritavancin (N=503) | Vancomycin (N=502)
Cellulitis (Infections and infestations) | 6 | 4
Osteomyelitis (Infections and infestations) | 4 | 0
Bronchitis (Infections and infestations) | 1 | 0
Gangrene (Infections and infestations) | 1 | 0
Infection (Infections and infestations) | 1 | 0
Necrotizing Fasciitis (Infections and infestations) | 1 | 0
Pneumonia (Infections and infestations) | 1 | 0
Wound Infection Staphylococcal (Infections and infestations) | 1 | 0
Cardiac Failure Congestive (Cardiac disorders) | 1 | 1
Electromechanical dissociation (Cardiac disorders) | 1 | 0
Mouth Ulceration (Gastrointestinal disorders) | 1 | 0
Rectal Hemorrhage (Gastrointestinal disorders) | 1 | 0
Hyperglycemia (Metabolism and nutrition disorders) | 1 | 0
Chest Pain (General disorders) | 1 | 0
Convulsion (Nervous system disorders) | 1 | 1
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 1 | 2
Angioedema (Skin and subcutaneous tissue disorders) | 1 | 0
Leukocytoplastic Vasculitis (Skin and subcutaneous tissue disorders) | 1 | 0
Tenosynovitis (Musculoskeletal and connective tissue disorders) | 1 | 0
Abscess Bacterial (Infections and infestations) | 0 | 1
Arthritis Bacterial (Infections and infestations) | 0 | 1
Extradural Abscess (Infections and infestations) | 0 | 1
Intervertebral Discitis (Infections and infestations) | 0 | 1
Lower Respiratory Tract Infection (Infections and infestations) | 0 | 1
Skin Bacterial Infection (Infections and infestations) | 0 | 1
Acute Myocardial Infarction (Cardiac disorders) | 0 | 2
Myocardial Ischaemia (Cardiac disorders) | 0 | 1
Constipation (Gastrointestinal disorders) | 0 | 1
Oesophagitis (Gastrointestinal disorders) | 0 | 1
Dehydration (Metabolism and nutrition disorders) | 0 | 1
Hyponatraemia (Metabolism and nutrition disorders) | 0 | 1
Metabolic Acidosis (Metabolism and nutrition disorders) | 0 | 1
Non-cardiac Chest Pain (General disorders) | 0 | 1
Headache (Nervous system disorders) | 0 | 1
Skin Ulcer (Skin and subcutaneous tissue disorders) | 0 | 1
Psychotic Disorder (Psychiatric disorders) | 0 | 1
Suicide Attempt (Psychiatric disorders) | 0 | 1
Anaphylactoid Reaction (Immune system disorders) | 0 | 1
Clavicle Fracture (Injury, poisoning and procedural complications) | 0 | 1
Renal Failure (Renal and urinary disorders) | 0 | 1
Skin Infection (Infections and infestations) | 0 | 2
Pyrexia (General disorders) | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 2% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Single-Dose 1200 mg Oritavancin (N=503) | Vancomycin (N=502)
nausea (Gastrointestinal disorders) | 45 | 60
headache (Nervous system disorders) | 35 | 28
vomiting (Gastrointestinal disorders) | 22 | 28
cellulitis (Infections and infestations) | 17 | 15
alanine aminotransferase increased (Investigations) | 16 | 10
infusion site phlebitis (General disorders) | 16 | 5
pyrexia (General disorders) | 15 | 11
infusion site extravasation (General disorders) | 15 | 10
tachycardia (Cardiac disorders) | 15 | 7
constipation (Gastrointestinal disorders) | 14 | 17
abscess limb (Infections and infestations) | 14 | 8
pruritus (Skin and subcutaneous tissue disorders) | 13 | 29
diarrhea (Gastrointestinal disorders) | 13 | 15
aspartate aminotransferase increased (Investigations) | 11 | 11
dizziness (Nervous system disorders) | 11 | 11

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes